CLINICAL TRIAL: NCT02151435
Title: Prospective Evaluation of Biomarker Profiles in Idiopathic Pulmonary Fibrosis
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Brown University (Other)
Responsible Party: Principal Investigator, Eric S. White, MD, Professor of Internal Medicine, University of Michigan
Other Study IDs: UM HUM00004076; R01HL109118 (NIH)
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: IPF
Keywords: Idiopathic Pulmonary Fibrosis; Biomarkers; Forced Vital Capacity; Diffusion Capacity for Carbon Monoxide; Prognosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood plasma obtained from individuals at 6-month intervals for up to 2 years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with IPF: Observation of longitudinal biomarkers in IPF patients

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a progressive, fatal, fibrotic disorder of the lung. The estimated prevalence is 30-80/100,000 in the United States with incidence estimates clearly rising. A major challenge in the care of patients with IPF is determining prognosis. The natural history of IPF is usually one of inexorable decline in lung function, ultimately resulting in death from respiratory failure. However, longitudinal physiologic decline in IPF is heterogeneous and difficult to predict in individual patients. While some patients with IPF may remain stable for years, in others the disease may progress rapidly over a relatively short time. We hypothesize that peripheral blood biomarkers based on extracellular matrix and matrix-modifying molecules will improve prognostication in patients with IPF.

ELIGIBILITY:
Inclusion Criteria:

1. Age 35-80 years, inclusive
2. Diagnosis of IPF by HRCT or surgical lung biopsy
3. Able to understand and provide informed consent

Exclusion Criteria:

1. AE-IPF during the prior year
2. Environmental exposure (occupational, drug, etc.) felt to be the etiology of the interstitial disease.
3. Diagnosis of collagen-vascular conditions according to published American College of Rheumatology criteria.
4. Significant airway obstruction (FEV1/FVC ratio < 0.60) or bronchodilator response, defined as a change in FEV1 ≥ 12% and absolute change > 200 mL OR change in FVC ≥ 12% and absolute change > 200 mL at baseline
5. Partial pressure of arterial oxygen (PaO2) < 55 mm Hg
6. Evidence of active infection
7. Listed for lung transplantation
8. Myocardial infarction, coronary artery bypass, or angioplasty within 6 months
9. Unstable angina pectoris or congestive heart failure requiring hospitalization or deteriorating within 6 months
10. Uncontrolled arrhythmia or hypertension
11. Known HIV, hepatitis C, cirrhosis, or chronic active hepatitis
12. Active substance and/or alcohol abuse
13. If you are pregnant or breastfeeding
14. Any condition other than IPF that is likely to result in your death within the next year
15. Any condition that, in the judgment of the PI, might cause participation in the study to be detrimental to you or that the PI deems makes you a poor candidate

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes subjects with IPF identified via the University of Michigan Interstitial Lung Disease Clinical-Radiologic-Pathologic Conference. The investigators will only enroll subjects in whom an IPF diagnosis is firmly established.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2013-08; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 1 year
  The primary outcome is your progression free survival as determined by time until any of: death, acute exacerbation of IPF, relative decline in FVC (liters) of at least 10% or DLCO (ml/min/mmHg) of 15% from baseline.

OTHER OUTCOMES:
Longitudinal change in biomarker levels | 1 year
  In exploratory analyses, longitudinal change in your biomarker expression will be correlated with your disease progression to determine if change in biomarker levels over time predict subsequent disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Eric S White, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Medical Center, Ann Arbor, Michigan, United States